CLINICAL TRIAL: NCT03765398
Title: Virtual-reality Based Cognitive-motor-balance (VR-CogMoBal) Training: Examining Behavioral and Neuromarkers for Fall-risk Reduction in Older Adults With Mild Cognitive Impairment
Brief Title: VR-CogMoBal Training for Reducing Falls Among Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tanvi Bhatt, Associate Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1257; 2P30AG022849-11 (NIH)
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Dual-task training; Virtual-reality exergaming; Cognitive-motor-balance training; Mild cognitive impairment; Older adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR Cognitive-motor-balance training (Experimental): Virtual reality based cognitive-motor balance (VR-CogMoBal) training will be delivered using the commercially available Wii-Fit Nintendo in conjunction with cognitive training. All participants will undergo 12 sessions of training in a tapering manner for four weeks with 90 minutes of training per session, i.e., 5 sessions for the first week, 3 sessions for the second week, and 2 sessions for the third and fourth week. Each session will be divided into 3 sub-sessions, where each sub-session will consist of playing 4 games in conjunction with cognitive task. All the games will be performed using a Wii-Fit balance board in front of a TV screen.
  Interventions: Behavioral: VR Cognitive-motor-balance training

INTERVENTIONS:
Behavioral: VR Cognitive-motor-balance training — The participant will play four of the six balance board games Table tilt, Tightrope, Soccer, Balance bubble, Light Run and Basic Step (each game is max 1.5 minutes). Each game will be superimposed with any 3 of the 6 cognitive tasks (word list generation consisting of verbal fluency (VF) and category fluency (CF), digit recall (DR), analogies (AN), mental arithmetic (MA), repeated letter (RL). The cognitive tasks will be randomized making sure that all the cognitive tasks are played with all the games. The cognitive and balance board game scores will be noted on the scoring sheet for each session. A total 10 minutes rest interval between every sub-session will be mandatorily provided.
  Other Names: VR-CogMoBal; Dual-task training

SUMMARY:
Older adults often display gait instability, impaired balance control and cognitive decline that lead to falls and fall risks. Approximately 60% of the elderly people with cognitive deficits experience a detrimental fall each year. Such motor and cognitive impairments further decreases physical activity levels in this population leading to restricted community integration, social behavior, depression and long-term disability. With the help of computer technology, studies have employed virtual-reality based interventions to address the above-mentioned concerns including sensori-motor, balance control and cognitive impairments. Previous studies have demonstrated promising results on improving the behavioral outcomes, and have identified such interventions have the potential to improve the underlying neurophysiological outcomes as well. While VR based training studies have demonstrated remarkable improvement in the balance control and gait parameters, physical activity levels and fall risk reduction, the gains on cognitive function is less pronounced. There is little evidence that VR-based training can explicitly address the higher executive cognitive domains associated with balance control and falls. Further, the effect of VR-based training on balance control and cognitive function is unknown among the older adults with mild cognitive impairment. Therefore, to address the cognitive domains explicitly, the current study aims to test the applicability of Wii-Fit Nintendo along with an additional cognitive load delivered via VR-based cognitive-motor training paradigm (VR-CogMoBal) in older adults with mild cognitive impairment. Lastly, the study also aims to identify the effect of such training on the underlying behavioral and neural outcomes. The behavioral outcomes will be assessed via performance on dual-tasking and clinical measures in the laboratory. The underlying neural outcomes will be assessed via fMRI outcomes. In order to determine the generalizing training effect at community level, a pilot sub-study to determine the physical activity levels post 4 weeks of training will also be conducted.

DETAILED DESCRIPTION:
Older adults suffer from mild cognitive impairments with a prevalence rate of 3% to 22% and an incidence rate of 1% to 6% per year in the United States. Along with age associated locomotor-balance impairments, such cognitive decline among the elderly is known to increase the risk of falls, reduced physical activity and community integration, thus contributing to long-term disability. Daily living activities comprises of several concurrent motor and cognitive performances (dual-tasking) such as shopping in a supermarket, that requires higher executive cognitive functions and intact locomotor-balance control abilities. Falls during dual-tasking occur mostly due to the interference caused, i.e. during dual-task performances, either one or both task (motor or cognitive) performance is deteriorated that is known as cognitive-motor interference. Given that dual-task performances decline due to age-associated factors, daily living activities are highly challenging and difficult to perform for older adults with mild cognitive impairment. Although there are several conventional methods that incorporate locomotor-balance training, the nature of such interventions does not result in pronounced cognitive gains. Additionally, these interventions lack multi-sensory feedback, and due to the monotonous and repeated task practice of exercises characteristic, individuals do not seem to adhere to therapy leading to less compliance and decreased motivation to exercise training. In order to overcome such barriers, alternate form of therapy with the help of Virtual-reality devices, especially off the shelf commercially available exercise platforms emerged for training purposes. Although there is evidence that VR based training improves locomotor-balance control and is known to implicitly address cognitive functions, there is no knowledge that such VR based training can explicitly address higher executive cognitive functions. Therefore, based on preliminary studies tested the efficacy of cognitive training along with exergaming delivered via the commercially available off the shelf device- Wii-fit Nintendo and demonstrated promising results in improving balance control and cognitive function among the individuals with Chronic Stroke. The study resulted in decreased cognitive-motor interference during dual-task performance thereby exhibiting an improved performance on both cognitive and balance control function. Currently, there is lack of knowledge in determining specific interventions for improving dual-task performances among the older adults with MCI. Given that mild cognitive impaired older adults suffer from both motor and cognitive impairments, there is a need for testing the feasibility of a similar intervention among them and determine the change in the underlying neural biomarkers.

Aim 1: The study is designed to test the feasibility (tolerability, compliance and effectiveness) of VR-CogMoBal training to improve physical function and reduce fall-risk in community-dwelling older adults with mild cognitive deficits by lowering cognitive-motor interference and dual task costs.

Hypothesis: Participants will tolerate the training paradigm and will demonstrate significant improvements in balance, gait, cardiovascular and cognitive performance under dual-task conditions.

Aim 2: To examine if the (VR-CogMoBal) will lead to higher cognitive function post-intervention.

Hypothesis: Post-training compared to pre-training participants will show significantly greater global cognitive function, executive and working memory and decreased cognitive-motor load.

Aim 3: To examine effect of VR-CogMoBal Training on changes in structural and functional connectivity within the cognitive-motor areas in the brain.

Hypothesis: Post-training compared to pre-training, participants will show increased structural and functional connectivity at rest in the default mode network (memory consolidation, self-referential memory), fronto-parietal and supplementary motor areas (motor planning and execution, attention).

Pilot Sub-study aim:

The study aims to monitor the change in the number of steps taken a day before undergoing VR training and 4 weeks post-training.

ELIGIBILITY:
Inclusion Criteria:

* MOCA less than 26 out of 30
* Bone density with a T-score ≥ -2.5
* Can understand and communicate in English
* Ability to stand for at least 5 minutes without an assistive device (length of a Wii Fit game)

Exclusion Criteria:

* any acute or chronic neurological (Stroke, Parkinson's disease, Alzheimer's disease), cardiopulmonary, musculoskeletal, or systemic diagnosis
* recent major surgery (< 6 months) or hospitalization (< 3 months)
* Use of any sedative drugs
* HR > 85% of age-predicted maximal heart rate (HRmax) (HRmax = 220 - age)
* systolic blood pressure (SBP) > 165 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg during resting), and/or oxygen saturation (measured by pulse oximeter) during resting < 90%
* Specific to MRI: Self-reported presence of pacemaker, metal implants, and/or Claustrophobia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi S Bhatt, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Baseline Measurements
Arm/Group | VR Cognitive-motor-balance Training
Started | 18
Completed | 14
Not Completed | 4
Period: Intervention
Arm/Group | VR Cognitive-motor-balance Training
Started | 14
Completed | 10
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale of 0-30] — The Montreal cognitive assessment scale measures the general cognitive function of an individual and includes domains of memory, executive function and information processing. The scale ranges from a minimum score of 0 to a maximum score of 30, higher score indicates better performance. We report the total score of the assessment scale. A score range from 26-30 indicates normal cognitive function, 19-25 indicates mild cognitive impairment, below 19 indicates dementia.
  units on a scale of 0-30 | 22.6 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Excursion
Description: It is the actual magnitude of a self-initiated movement (i.e., how far did he/she actually reach a target) without taking a step or losing balance measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 5)
Measure: Mean (Standard Deviation); unit: percentage of center of pressure motion
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 10
percentage of center of pressure motion
  Maximum excursion in forward Direction, Pre-Training | 80.9 (13.8)
  Maximum excursion in Forward Direction, Post-Training | 86.5 (15)
  Maximum excursion in Backward Direction, Pre-Training | 66.8 (17.7)
  Maximum excursion in Backward Direction, Post-Training | 80.9 (11.8)
  Maximum excursion in Left Direction, Pre-Training | 80.7 (11.0)
  Maximum excursion in Left Direction, Post-Training | 87.1 (5.3)
  Maximum excursion in Right Direction, Pre-Training | 76.4 (11.2)
  Maximum excursion in Right Direction, Post-Training | 87.3 (6.9)
  Maximum excursion in Forward Direction while performing auditory clock test, Pre-Training | 72.0 (23.6)
  Maximum excursion in Forward Direction while performing auditory clock test, Post-Training | 84.2 (17.4)
  Maximum excursion in Backward Direction while performing auditory clock test, Pre-Training | 61.9 (15.1)
  Maximum excursion in Backward Direction while performing auditory clock test, Post-Training | 66.2 (21.1)
  Maximum excursion in Left Direction while performing auditory clock test, Pre-Training | 71.8 (14.2)
  Maximum excursion in Left Direction while performing auditory clock test, Post-Training | 84.7 (6.8)
  Maximum excursion in Right Direction while performing auditory clock test, Pre-Training | 72.9 (14.2)
  Maximum excursion in Right Direction while performing auditory clock test, Post-Training | 86.1 (9.2)
  Maximum excursion in Forward Direction while performing letter number sequencing, Pre-Training | 69.6 (20.5)
  Maximum excursion in Forward Direction while performing letter number sequencing, Post-Training | 80.7 (16.9)
  Maximum excursion in Backward Direction while performing letter number sequencing, Pre-Training | 58.1 (21.4)
  Maximum excursion in Backward Direction while performing letter number sequencing, Post-Training | 71.2 (16.3)
  Maximum excursion in Left Direction while performing letter number sequencing, Pre-Training | 68.2 (18.0)
  Maximum excursion in Left Direction while performing letter number sequencing, Post-Training | 84.8 (5.8)
  Maximum excursion in Right Direction while performing letter number sequencing, Pre-Training | 72.9 (14.0)
  Maximum excursion in Right Direction while performing letter number sequencing, Post-Training | 80.3 (10.2)

2. Primary Outcome: Change in 4 Meter Walk Test
Description: The total time taken to complete the 4 meters will be noted. Speed will then be determined by using the formula distance (4 meters) covered by time taken to complete the test. Higher speed indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 5)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 10
m/s
  Pre-Training | 0.95 (0.08)
  Post-Training | 1.08 (0.14)

3. Primary Outcome: Change of Accuracy in Letter Number Sequencing
Description: This is an oral trail making test which includes listing alternate letter and number from the cue given in sequence. This test will be performed under single and dual-task conditions.
  For the auditory clock test, the participant is provided with cues that include different times of the day (e.g., 3.15) and the participant has to answer a yes if the hour and the minute hand of the clock are on the same side and no if the hour and minute hand are on opposite side of the clock.
  For the letter number sequencing test, the participant will be provided sets of letters and numbers (e.g.., A1) and will be asked to list in sequence the consecutive letter and numbers (e.g., B2, C3, D4, E5) until the next cue is provided.
  The performance will be measured in terms of accuracy (number of correct responses out of the total responses) for both the tests. Higher accuracy i.e., higher percentage indicates better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 5)
Measure: Mean (Standard Deviation); unit: percentage of total responses
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 10
percentage of total responses
  Single Task, Pre-Training | 65 (27)
  Single Task, Post-Training | 77 (19)
  Dual Task during forward leaning, Pre-Training | 69 (23)
  Dual Task during forward leaning, Post-Training | 63 (33)
  Dual Task during backward leaning, Pre-Training | 40 (38)
  Dual Task during backward leaning, Post-Training | 51 (30)
  Dual Task during left leaning, Pre-Training | 51 (30)
  Dual Task during left leaning, Post-Training | 57 (31)
  Dual Task during right leaning, Pre-Training | 50 (31)
  Dual Task during right leaning, Post-Training | 64 (30)

4. Primary Outcome: Change in Working Memory
Description: List Sorting Memory test to evaluate working memory. This test requires the participant to recall and sequentially list the visually and orally presented stimuli. The accuracy of the participants response is computer generated. Higher value indicate better performance. The total possible responses are 28.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 5)
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 10
correct responses
  Pre-Training | 12.1 (1.0)
  Post-Training | 13.6 (2.8)

5. Primary Outcome: Change in Episodic Memory
Description: Picture sequence memory test will assess episodic memory of the individual. The number of adjacent pairs of pictures placed correctly will score a point. The scores are computer generated. Higher value indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 5)
Measure: Mean (Standard Deviation); unit: accuracy (%)
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 10
accuracy (%)
  Pre-Training | 17.3 (9.6)
  Post-Training | 27.4 (9.1)

6. Primary Outcome: Change in Accuracy of Flanker Inhibitory Control and Attention Test
Description: Flanker inhibitory control and attention test is used to evaluate the participants ability to inhibit the attention to the stimulus flanking it and focus on a particular stimulus. Accuracy of the responses are recorded and the scores are computer generated. Higher value indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 5)
Measure: Mean (Standard Deviation); unit: % accurate
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 10
% accurate
  Pre-Training | 39.6 (0.97)
  Post-Training | 40 (0.0)

7. Primary Outcome: Change in Cognitive Flexibility and Attention
Description: Dimensional Change card sort assesses cognitive flexibility and attention. Participants are asked to match a series of bivalent pictures either by colors or shapes accordingly. Responses are computer recorded and accuracy scores are computer generated. Higher value indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 5)
Measure: Mean (Standard Deviation); unit: % accurate
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 10
% accurate
  Pre-Training | 34.3 (5.4)
  Post-Training | 38.5 (3.7)

8. Primary Outcome: Change in Processing Speed
Description: Pattern comparison processing speed test is used to evaluate the processing speed. The participants are expected to respond whether the two pictures side-by side are same or not the same. Accuracy will be recorded by the number of correct responses out of the total questions in 90 seconds. Scores are computer generated. Higher value indicate better performance.
Time Frame: Baseline (Week 0) and Immediate Post-training (Week 5)
Measure: Mean (Standard Deviation); unit: percentage of accurate responses
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 10
percentage of accurate responses
  Pre-Training | 26.4 (4.2)
  Post-Training | 29.2 (5.5)

9. Secondary Outcome: Change in Movement Velocity
Description: It is the average speed of center of gravity movement during intentional movement measured in degrees per second under single and dual-task conditions. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Immediate post-training (Week 5)
Population: Due to the emergence of the COVID-19 pandemic, this study was conducted primarily on Zoom, preventing the collection of data for this outcome measure, as the assessment is typically conducted in person.
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

10. Secondary Outcome: Changes in End Point Excursion
Description: It is the magnitude of a self-initiated movement (i.e., how far he/she wills to reach a target) without taking a step or losing balance measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Directional Control
Description: It is the quality of a self-initiated movement (i.e., amount of movement actually exhibited towards the target to the amount of extraneous movement away from the target) measured in percentage under single and dual-task conditions. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Postural Stability During Reactive Balance Control (Single and Dual-task)
Description: Reactive balance control will be examined via the stance perturbation test under single and dual-task conditions (simultaneous performance of Letter number sequencing task or auditory stroop task). Postural stability can be defined as simultaneous control of center of mass (COM) position and velocity during slip-like or trip like perturbation relative to the rear edge of base of support (rear heel). The position is normalized with the individual's foot length, and velocity by square root of gravitational acceleration and individual's body height. Larger values indicate greater stability.
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in Accuracy of Auditory Stroop
Description: This test involves responding to the pitch (high or low) of the words "High" or "Low". This test will be performed under single and dual-task conditions.
  Accuracy (number of correct responses out of the total responses) of Auditory stroop will be calculated. Higher accuracy indicates better performance. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

14. Secondary Outcome: Change in Dual-task Cost
Description: Dual-task motor and cognitive cost will be calculated using the formula- [(Dual-task performance- Single Task performance)/Single task performance*100]. This will be calculated for dual-task performance during intentional postural sway, reactive balance control and gait conditions. Lower cost indicates better performance.
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in Gait Parameters
Description: Spatial and temporal gait parameters like step length, cadence and stride length will be determined during single and dual-task walking performance via the GaitRite mat. Higher values for step length and stride length, and lower cadence indicates better performance.
Time Frame: Baseline (Week 0) and post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

16. Secondary Outcome: Change in Interference in the Reaction Time
Description: Interference in the reaction time via visual stroop task where the individual is expected to respond to the color in which the word is printed and not read the word. Performance will be identified via time taken to complete the test. Lower time indicates better performance.
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

17. Secondary Outcome: Change in Language Fluency
Description: Language fluency via verbal and category task will be administered. Performance will be identified via the total number of appropriate words responded on each of the task. Higher values indicate better performance.
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

18. Secondary Outcome: Change in Interference in Reaction Time
Description: The individual is asked to hit a key on the number keypad when a cue appears on the screen. Performance will be identified with time taken to hit the key after the individual sees the cue in seconds. Lower time indicates better performance.
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

19. Secondary Outcome: Change in Paired Associative Learning
Description: Paired associated learning via grid task will be administered. Accuracy (number of correct responses out of the total responses) will be represented in percentage. Higher value indicates better performance.
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

20. Secondary Outcome: Change in Spatial Working Memory
Description: List Sorting Memory test to evaluate working memory. This test requires the participant to recall and sequentially list the visually and orally presented stimuli. The accuracy of the participant's response is computer generated. Higher value indicates better performance. The minimum score is 0% and maximum score is 100%
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

21. Secondary Outcome: Change in Reaction Time
Description: as for outcome 18
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

22. Secondary Outcome: Changes in Fractional Anisotropy
Description: Fractional anisotropy (FA) is a scalar measure derived from diffusion tensor imaging (DTI) that quantifies the directional dependence of water molecule diffusion in biological tissues. Ranging from 0 (completely isotropic diffusion, as in cerebrospinal fluid) to 1 (fully anisotropic diffusion, seen in highly organized white matter tracts), FA reflects microstructural properties such as axonal density, myelination, and fiber coherence. Higher values indicate better integrity of white matter tracts
Time Frame: Baseline (Week 0) and Post-training (Week 4)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

23. Secondary Outcome: Berg Balance Scale
Description: The Berg Balance Scale (BBS) is a standardized clinical assessment tool designed to evaluate static and dynamic balance abilities, primarily in older adults and individuals with neurological conditions. The scale score ranges form a minimum of 0 to a maximum of 56, with higher scores indicating better balance performance
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

24. Secondary Outcome: Change in Physical Activity Level (Questionnaires)
Description: The Physical Activity Scale for the Elderly (PASE) is a validated self-report questionnaire designed to quantify physical activity levels in adults aged 65+ through occupational, household, and leisure activities over a 7-day period. The scores ranges from 0-793 with higher score indicating better performance.
Time Frame: Baseline (Week 0) and Post-training (Week 5)
Population: as for outcome 9
Arm/Group | VR Cognitive-motor-balance Training
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 month during training and during the pre-training and post-training session
Arm/Group | VR Cognitive-motor-balance Training
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT03765398/Prot_SAP_000.pdf